CLINICAL TRIAL: NCT00190710
Title: A Randomized Phase III Trial of Paraplatin (Carboplatin) + Gemzar Versus Gemzar Alone in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: A Trial of Carboplatin and Gemcitabine Versus Gemcitabine Alone in Patients With Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9297; B9E-US-S358
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Carboplatin

INTERVENTIONS:
Drug: Gemcitabine
Drug: Carboplatin

SUMMARY:
To determine and compare the median survival produced by combined Gemcitabine plus Paraplatin versus Gemcitabine as a single-agent in patients with NSCLC and a PS equal to 2.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic new diagnosis of NSCLC, Stage IIIB with a cytologically positive pleural or pericardial effusion or Stage IV.
* No prior chemotherapy, including adjuvant or neoadjuvant therapy, for the treatment of NSCLC.
* ECOG Performance Status of 2 .
* Patients must be at least 3 weeks since major surgery. Patients must be at least 1 week since surgery, such as mediastinoscopy, pleuroscopy, or thoracostomy.
* Patients must have measurable disease, defined as lesions that can be accurately measured in at least 1 dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than 10 mm with spiral CT scan.

Exclusion Criteria:

* Any prior radiation therapy to the thoracic area.
* Active and ongoing systemic infection.
* Prior radiation to greater than 25% of the bone marrow.
* ECOG PS other than 2
* Patients with a known hypersensitivity to gemcitabine and carboplatin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242
Dates: Start 2004-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To determine and compare the median survival produced by combined Gemcitabine plus Paraplatin versus Gemcitabine as a single-agent in patients with NSCLC and a PS equal to 2.

SECONDARY OUTCOMES:
To determine and compare the 1-year survival produced by combined Paraplatin (carboplatin) + Gemcitabine versus Gemcitabine as a single-agent in patients with NSCLC and a PS equal to 2
To determine the safety of combined Gemcitabine plus Paraplatin versus Gemcitabine as a single-agent in patients with NSCLC and a PS equal to 2
To compare the response rate between treatment groups
To compare the changes in QOL between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

REFERENCES:
- [Derived] Gijtenbeek RG, de Jong K, Venmans BJ, van Vollenhoven FH, Ten Brinke A, Van der Wekken AJ, van Geffen WH. Best first-line therapy for people with advanced non-small cell lung cancer, performance status 2 without a targetable mutation or with an unknown mutation status. Cochrane Database Syst Rev. 2023 Jul 7;7(7):CD013382. doi: 10.1002/14651858.CD013382.pub2. PMID 37419867
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com